CLINICAL TRIAL: NCT01896921
Title: Switch to Maraviroc and Integrase Strand Transfer Inhibitor Combination Therapy (a Triple Class-Sparing Regimen) for the Treatment of HIV-1-Infected Patients on Suppressive Antiretroviral Regimens
Brief Title: Switch to Maraviroc + Integrase Inhibitor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, David Riedel, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00056162
Record Dates: First submitted 2013-06-27; First posted 2013-07-11 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — Raltegravir Potassium; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc + Raltegravir or Dolutegravir (Experimental): Maraviroc 300 mg tablet twice a day plus Raltegravir 400 mg tablet twice a day or Dolutegravir 50 mg tablet once a day for 48 weeks
  Interventions: Drug: Switch to Maraviroc + Raltegravir or Dolutegravir

INTERVENTIONS:
Drug: Switch to Maraviroc + Raltegravir or Dolutegravir — Change HIV-infected patients on stable, suppressed ART regimens for at least 1 year to experimental regimen of Maraviroc + Raltegravir or Dolutegravir for 48 weeks

SUMMARY:
This clinical study proposes to evaluate the combination of maraviroc with an integrase strand transfer inhibitor (either raltegravir or dolutegravir) in antiretroviral-experienced patients to document the efficacy, safety, and tolerability of this combination in order to provide clinicians with a treatment regimen that minimizes the risk of metabolic complications by avoidance of NRTI/NNRTIs and PIs. The development of an alternative ART regimen which lessens the risk of metabolic complications could improve long-term adherence and reduce the risk of certain co-morbidities associated with long-term ART use. If this new combination is found to be as efficacious as the standard regimen with enhanced tolerability and improved metabolic effects, there is great potential for altering the current practice of HIV medicine.

DETAILED DESCRIPTION:
Description of the study design:

The study will enroll 30 HIV-infected patients on a stable ART regimen with a suppressed HIV RNA < 50 copies/ml for at least one year. Patients will be switched to the experimental regimen (maraviroc 300 mg twice a day plus either raltegravir 400 mg twice a day or dolutegravir 50 mg once a-day) and followed for 96 weeks. The decision to use raltegravir or dolutegravir will be left to investigator/subject preference, as the two integrate inhibitors are largely interchangeable aside from twice daily (raltegravir) vs. daily (dolutegravir) dosing.

Primary endpoint:

* The primary endpoint is the proportion of patients virologically suppressed (HIV RNA < 50 copies/ml) at 48 weeks.

Definitions:

* Virologic suppression is an HIV RNA < 50 copies/ml.
* Virologic failure is an HIV RNA ≥ 50 copies/ml confirmed on 2 separate occasions, separated by > 1 week after viral suppression.

Secondary endpoints:

* The percent change in total cholesterol, LDL, and HDL at 48 and 96 weeks.
* The number of adverse events.
* The proportion of patients who are virologically suppressed (HIV RNA < 50 copies/ml) at 96 weeks.

Exploratory endpoints:

* Telomerase activity and telomere length measured at baseline and 24, 48, and 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age between 18 and 75 years
* CD4 count nadir ≥ 250 cells/mm3
* HIV RNA ≤ 50 copies/ml for ≥ 12 months while taking any ART regimen

  o One virologic blip ≤ 400 copies/ml permissible within the 12 months
* CCR5 tropic virus as defined by:

  * trofile/tropism testing if available, OR
  * DNA trofile if no trofile/tropism test available and CD4 nadir 250-499 cells/mm3, OR
  * CD4 nadir ≥ 500 cells/mm3

Exclusion Criteria:

* Age < 18 or > 75 years
* CD4 count nadir < 250 cells/mm3
* Dual/mixed or X4 tropic virus if tested prior to viral suppression or if performed by DNA trofile testing at any time
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limits of normal
* Women who:

  * are currently pregnant or breastfeeding
  * are of child-bearing age and do not agree to remain abstinent or use (or have their partner use) an acceptable method of birth control throughout the study. Acceptable method of birth control is defined as intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, vasectomy.
* History of any malignancy except non-melanoma skin cancer
* Concomitant use of drugs known to impact or be impacted in terms of pharmacokinetics or drug-drug interactions with either raltegravir or maraviroc. This includes:

  * Inducers of UGT1A1 (such as rifampin, phenytoin, phenobarbital rifabutin, St. John's wort)
  * CYP3A inhibitors (such as ketoconazole, itraconazole, clarithromycin, nefazodone, and telithromycin)
  * CYP3A inducers (such as rifampin, carbamazepine, phenobarbital and phenytoin)
* Subject requires or is anticipated to require any of the prohibited medications noted in the protocol
* Enrollment in an experimental protocol having received investigational agents (antiretroviral or non-antiretroviral) within 30 days of study enrollment
* Chronic active hepatitis B infection as defined by presence of HBsAg
* Subject has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate.
* Subject is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Riedel, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maraviroc + Raltegravir or Dolutegravir
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc + Raltegravir or Dolutegravir
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [54 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Virologically Suppressed (HIV RNA <50 Copies/ml) at 48 Weeks.
Description: Number of patients virologically suppressed (HIV RNA <50 copies/ml) at 48 weeks.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc + Raltegravir or Dolutegravir
Number analyzed (Participants) | 7
Participants | 5

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events
Time Frame: 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc + Raltegravir or Dolutegravir
Number analyzed (Participants) | 7
Participants | 3

3. Secondary Outcome: Number of Patients Who Are Virologically Suppressed (HIV RNA < 50 Copies/ml)
Description: Number of patients who are virologically suppressed (HIV RNA < 50 copies/ml)
Time Frame: 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc + Raltegravir or Dolutegravir
Number analyzed (Participants) | 7
Participants | 4

ADVERSE EVENTS:
Time Frame: 96 weeks
Arm/Group | Maraviroc + Raltegravir or Dolutegravir
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc + Raltegravir or Dolutegravir (N=7)
Hyperglycemia (Endocrine disorders) | 1 (1)
Mechanical fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT01896921/Prot_SAP_000.pdf